CLINICAL TRIAL: NCT02169219
Title: Short-Course Glucocorticoids and Rituximab in ANCA-Associated Vasculitis
Brief Title: Pilot Study of Short-Course Glucocorticoids and Rituximab for Treatment of ANCA-Associated Vasculitis
Acronym: SCOUT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Stone, John H, M.D., M.P.H, Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012P001427
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Granulomatosis With Polyangiitis; Microscopic Polyangiitis
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis | interventions — Glucocorticoids; Prednisone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Glucocorticoids and Rituximab (Experimental): This is a single-arm trial. All patients receive both rituximab and glucocorticoids. The protocol calls for the discontinuation of prednisone within two months of the baseline visit.
  Interventions: Drug: Glucocorticoids; Drug: Rituximab

INTERVENTIONS:
Drug: Glucocorticoids — Patients will begin prednisone therapy at a dose selected by the investigator or the treating physician with oral prednisone 60mg or 1mg/kg (if weight less than 60kg) or intravenous methylprednisolone, up to 1g/day for three days.
  Prednisone will be tapered over 8 weeks as follows:
  * 60mg for 2 weeks
  * 40mg for 2 weeks
  * 30mg for 1 week
  * 20mg for 1 week
  * 10mg for 1 week
  * 5mg for 1 week
  Other Names: Prednisone
Drug: Rituximab — Rituximab will be administered in four weekly doses at 375mg/m2
  Other Names: Rituxan

SUMMARY:
The purpose of this pilot study is to test whether an 8-week course of glucocorticoids, combined with rituximab, is effective in treating ANCA-associated vasculitis.

DETAILED DESCRIPTION:
The primary aim of this pilot study is to examine whether an 8 week course of glucocorticoids, in combination with rituximab, is effective in inducing and maintaining disease remission for up to 6 months in a subset of patients with ANCA-associated vasculitis (AAV) who have a more favorable prognosis.

This pilot study will enroll 20 patients with active AAV. Close patient follow-up will insure that any patients who require courses of glucocorticoids longer than two months will receive longer therapy, if appropriate for their well-being.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 18-85 years old
* Diagnosis of GPA or MPA according to the definitions of the Chapel Hill Consensus Conference
* New diagnosis or disease flare with a Birmingham Vasculitis Activity Score/Wegener's granulomatosis (BVAS/WG) of > 3

Exclusion Criteria:

* Renal disease in patients with PR3-ANCA as defined by any of the following:
* Urinary red blood cell casts
* Biopsy-proven glomerulonephritis
* Increase in serum creatinine of >30% over baseline
* Severe renal disease in patients with MPO-ANCA as defined by both of the following:
* Urinary red blood cell casts or biopsy-proven glomerulonephritis
* Estimated glomerular filtration rate < 30 ml/min/1.73m2
* Diffuse alveolar hemorrhage requiring ventilatory support
* GC treatment for longer than 14 days prior to enrollment unless patient has been on a stable maintenance dose of prednisone at the time of the flare
* Daily oral cyclophosphamide within 1 month prior to enrollment
* Completed a remission induction course of cyclophosphamide or rituximab within 4 months of enrollment
* Hepatitis B infection
* HIV infection
* History of anti-GBM disease
* Other uncontrolled disease, including drug and alcohol abuse, that may interfere with the study
* Pregnancy or breastfeeding
* History of severe allergic reactions to human or chimeric monoclonal antibodies

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2016-08-17 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H Stone, MD, Principal Investigator — Massachusetts General Hospital and Harvard Medical School
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon request - without personal health information - following completion of the analysis. Inquiries should be directed to the Principal Investigator.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * New diagnosis or flare of previously diagnosed disease in patients followed in the Massachusetts General Hospital (MGH) Rheumatology or Nephrology Units.
  * New diagnosis or flare of previously diagnosed disease in patients hospitalized at MGH.
Groups:
- Glucocorticoids and Rituximab: All patients receive both rituximab and glucocorticoids. The protocol calls for the discontinuation of prednisone within two months of the baseline visit.
Period: Overall Study
Arm/Group | Glucocorticoids and Rituximab
Started | 20
Completed | 14
Not Completed | 6
Not completed — Lack of Efficacy | 6

BASELINE CHARACTERISTICS:
Groups:
- Glucocorticoids and Rituximab: This is a single-arm trial. All patients receive both rituximab and glucocorticoids. The protocol calls for the discontinuation of prednisone within two months of the baseline visit.
  Glucocorticoids: Patients will begin prednisone therapy at a dose selected by the investigator or the treating physician with oral prednisone 60mg or 1mg/kg (if weight less than 60kg) or intravenous methylprednisolone, up to 1g/day for three days.
  Prednisone will be tapered over 8 weeks as follows:
  * 60mg for 2 weeks
  * 40mg for 2 weeks
  * 30mg for 1 week
  * 20mg for 1 week
  * 10mg for 1 week
  * 5mg for 1 week
  Rituximab: Rituximab will be administered in four weekly doses at 375mg/m2
Arm/Group | Glucocorticoids and Rituximab
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Birmingham Vasculitis Activity Score for Wegener's Granulomatosis(BVAS/WG) [Mean (Full Range); unit: units on a scale] — Birmingham Vasculitis Activity Score for Wegener's Granulomatosis(BVAS/WG, range 0-64). The total score is composed of 34 predefined items, units on a scale, grouped into 9 organ systems. Each item carries a weight from 1-3, depending on disease severity. Subjects with a score of 3 or higher were invited to participate in the trial. A score of 0 indicates no disease activity; a higher score indicates worsening disease.
  units on a scale | 5 [3 to 11]
Disease group [Count of Participants; unit: Participants] — Disease type (GPA or MPA)
  Participants
    Granulomatosis with polyangiitis (GPA) | 14
    Microscopic polyangiitis (MPA) | 6
    Indeterminate | 0
anti-neutrophil cytoplasmic antibody (ANCA) [Count of Participants; unit: Participants] — ANCA type and titer were determined by ELISA.
  Participants
    myeloperoxidase (MPO) | 11
    proteinase (PR3) | 7
    Negative | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission
Description: We examined whether an 8-week glucocorticoid course in combination with rituximab (RTX) would induce disease remission in patients with AAV. The primary outcome was disease remission off steroids at 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Glucocorticoids and Rituximab: Glucocorticoids: Patients will begin prednisone therapy at a dose selected by the investigator or the treating physician with oral prednisone 60mg or 1mg/kg (if weight less than 60kg) or intravenous methylprednisolone, up to 1g/day for three days.
  Prednisone will be tapered over 8 weeks as follows:
  * 60mg for 2 weeks
  * 40mg for 2 weeks
  * 30mg for 1 week
  * 20mg for 1 week
  * 10mg for 1 week
  * 5mg for 1 week
  Rituximab will be administered in four weekly doses at 375mg/m2
Arm/Group | Glucocorticoids and Rituximab
Number analyzed (Participants) | 20
Participants | 14

2. Secondary Outcome: Disease Response
Description: Number of patients achieving disease response defined as, no new disease manifestations; no worsening of existing disease; stable or improved BVAS/WG score at 4 weeks.
Time Frame: 4 weeks
Population: Number of patients having a disease response
Measure: Count of Participants; unit: Participants
Groups:
- Rituximab and Glucocorticoids: Prednisone will be tapered over 8 weeks as follows:
  * 60mg for 2 weeks
  * 40mg for 2 weeks
  * 30mg for 1 week
  * 20mg for 1 week
  * 10mg for 1 week
  * 5mg for 1 week
  Rituximab administered in 4 weekly doses at 375 mg/m2
Arm/Group | Rituximab and Glucocorticoids
Number analyzed (Participants) | 20
Participants | 20

3. Secondary Outcome: Partial Remission
Description: Number of patients entering partial remission, defined as no new disease manifestations, no worsening of existing disease and BVAS/WG < 3.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Glucocorticoids and Rituximab
Number analyzed (Participants) | 20
Participants | 20

4. Secondary Outcome: Sustained Complete Remission
Description: Number of patients entering sustained remission defined as BVAS/WG = 0, prednisone dose = 0 and no disease flares during the study period.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Glucocorticoids and Rituximab
Number analyzed (Participants) | 20
Participants | 14

5. Secondary Outcome: Limited Flares
Description: Number of limited flares defined as a new occurrence or worsening of one or more minor BVAS/WG items and a total BVAS/WG ≤ 3
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Glucocorticoids and Rituximab: Glucocorticoids: Patients will begin prednisone therapy at a dose selected by the investigator or the treating physician with oral prednisone 60mg or 1mg/kg (if weight less than 60kg) or intravenous methylprednisolone, up to 1g/day for three days.
  Prednisone will be tapered over 8 weeks as follows:
  * 60mg for 2 weeks
  * 40mg for 2 weeks
  * 30mg for 1 week
  * 20mg for 1 week
  * 10mg for 1 week
  * 5mg for 1 week
  Rituximab: Rituximab will be administered in four weekly doses at 375mg/m2
Arm/Group | Glucocorticoids and Rituximab
Number analyzed (Participants) | 20
Participants | 2

6. Secondary Outcome: Severe Flares
Description: Number of severe flares defined as flare with BVAS/WG > 3 or experiencing one of the major BVAS/WG items
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Glucocorticoids and Rituximab
Number analyzed (Participants) | 20
Participants | 5

7. Secondary Outcome: Early Treatment Failures
Description: Number of early treatment failures defined as patients who have new or worsening disease manifestations assessed at 4 weeks after study entry
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Glucocorticoids and Rituximab
Number analyzed (Participants) | 20
Participants | 0

8. Secondary Outcome: Vasculitis Damage Index (VDI)
Description: The Vasculitis Damage Index (VDI) is a single-page catalog of damage items separated into 11 groupings of items by organ system. There are a total of 60 items. Each item is recorded if it occurred since the onset of vasculitis, has been present for at least 3 months, or occurred at least 3 months ago. Each item of damage is scored as present (1) or absent (0), yielding a maximum score of 60.
Time Frame: 24 months
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Groups:
- Glucocorticoids and Rituximab: Measure Description: Disease damage was assessed by the Vasculitis Damage Index (VDI) at baseline and end of study
Arm/Group | Glucocorticoids and Rituximab
Number analyzed (Participants) | 20
units on a scale
  Baseline VDI score | 0 [0 to 1]
  24 month VDI score | 0.5 [0 to 2]

ADVERSE EVENTS:
Time Frame: Reports of unanticipated problems involving risks to subjects or others are to be submitted to the IRB within 5 working days/7 calendar days of the date the investigator first becomes aware of the problem. Adverse events were collected through the 6 month study duration.
Description: Serious adverse event means any event temporally associated with the subject's participation in research that meets any of the following criteria:
  1) hospitalization or prolonged hospitalization 2.)One severe flare - defined as BVAS/WG ≥ 3 or experiencing one of the major BVAS/WG items) 3.) unexpected and related to the investigation drug
Groups:
- Glucocorticoids and Rituximab: Patients will begin prednisone therapy at a dose selected by the investigator or the treating physician with oral prednisone 60mg or 1mg/kg (if weight less than 60kg) or intravenous methylprednisolone, up to 1g/day for three days.
  Prednisone will be tapered over 8 weeks as follows:
  * 60mg for 2 weeks
  * 40mg for 2 weeks
  * 30mg for 1 week
  * 20mg for 1 week
  * 10mg for 1 week
  * 5mg for 1 week
  Rituximab: Rituximab will be administered in four weekly doses at 375mg/m2
Arm/Group | Glucocorticoids and Rituximab
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 11/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glucocorticoids and Rituximab (N=20)
Severe flares (Immune system disorders) | 5 (5)
myocardial infarction (Cardiac disorders) | 1 (1)
atrial fibrillation, (Cardiac disorders) | 1 (1)
syncope (Immune system disorders) | 1 (1)
Thyroid maligancy (Endocrine disorders) | 2 (2)
Uterine malignancy (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT02169219/Prot_SAP_000.pdf